CLINICAL TRIAL: NCT00928096
Title: Breathing Adapted Radiotherapy for Mediastinal Lymphoma
Status: Completed | Type: Observational
Sponsor: Peter Meidahl Petersen (Other)
Collaborators: University of Copenhagen (Other)
Responsible Party: Sponsor-Investigator, Peter Meidahl Petersen, MD.Ph.D, Rigshospitalet, Denmark, Rigshospitalet, Denmark
Organization: Rigshospitalet, Denmark (Other)
Other Study IDs: HN-gating-001; H-D-2007-0069
Record Dates: First submitted 2009-06-23; First posted 2009-06-25 (Estimated); Last update posted 2014-10-21 (Estimated); Status verified 2014-10

CONDITIONS: Lymphoma
Keywords: Lymphoma; Radiotherapy; Positron-Emission Tomography; CT scan
MeSH Terms: conditions — Lymphoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
In this study, radiation therapy plans will be made for 20 consecutive patients with mediastinal Hodgkin lymphoma or aggressive non-Hodgkin lymphoma. One plan is done using a breathing adapted pre-chemo PET-CT scan fused with a post-chemo planning CT scan and another plan is done using the standard procedure with pre-chemo PET-CT fused with post-chemo planning CT scan. Dose levels to the lymphoma and to the organs of risk will be compared in each patient. The best radiation therapy plan will be used to treat the patient.

DETAILED DESCRIPTION:
Radiotherapy using a breathing adapted therapy scan is a routine technique in breast cancer. Breathing adapted radiotherapy may also reduce radiation dose to organs at risk, e.g. heart and lung, in patients with mediastinal Hodgkin lymphoma and aggressive non-Hodgkin lymphomas.

Optimal radiation therapy of these lymphoma patients includes radiotherapy planning using pre-chemotherapy PET-scanning, fused with a post-chemo planning CT-scan. This makes accurate treatment of pre-chemo involved volume possible and also accurate radiation of the post-chemo involved volume possible. Thus, the optimal breathing adapted radiation requires planning using a breathing adapted pre-chemo PET-CT scan fused with a breathing adapted post-chemo planning CT scan. In this study, 20 consecutive patients with mediastinal Hodgkin lymphoma and aggressive non-Hodgkin lymphomas will have combination therapy with chemotherapy and radiation therapy to involved nodes. Two radiation therapy plans will be made for each patient: one using a breathing adapted pre-chemo PET-CT scan fused with a post-chemo planning CT scan, and one using the standard procedure of a pre-chemo PET-CT scan fused with post-chemo planning CT scan. Dose levels to the lymphoma and to the organs of risk will be compared in each patient. The best radiation therapy plan will be used to treat the patient.

ELIGIBILITY:
Inclusion Criteria:

* Stage I/II mediastinal Hodgkin lymphoma or aggressive non-Hodgkin lymphomas
* Treatment plan includes radiotherapy

Exclusion Criteria:

* Not able to comply to breathing adapted therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 20 consecutive patients with mediastinal Hodgkin lymphoma and aggressive non-Hodgkin lymphomas refered to Hematological Clinic, Copenhagen University Hospital, Rigshospitalet
Sampling Method: Non-Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2009-06; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Estimated radiation dose levels to the lymphoma and to the organs of risk | Before day 1 of radiation therapy

CONTACTS AND LOCATIONS:
Overall Officials: Peter M Petersen, MD, Ph.D, Principal Investigator — Rigshospitalet, Denmark
Locations (1):
- Department of Hematology and Department of Radiation Oncology, Copenhagen University Hospital, Rigshospitalet, Copenhagen, Denmark

REFERENCES:
- [Result] Petersen PM, Aznar MC, Berthelsen AK, Loft A, Schut DA, Maraldo M, Josipovic M, Klausen TL, Andersen FL, Specht L. Prospective phase II trial of image-guided radiotherapy in Hodgkin lymphoma: benefit of deep inspiration breath-hold. Acta Oncol. 2015 Jan;54(1):60-6. doi: 10.3109/0284186X.2014.932435. Epub 2014 Jul 15. PMID 25025999